CLINICAL TRIAL: NCT06321016
Title: POZIKIDS: Exercise and Comprehensive Care to Improve the Quality of Life of Children and Adolescents With Cancer
Acronym: PoziKids
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nere Mendizabal (Other Government)
Responsible Party: Sponsor-Investigator, Nere Mendizabal, Nurse, Basque Health Service
Organization: Basque Health Service (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023111039
Record Dates: First submitted 2024-02-06; First posted 2024-03-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Exercise; Childhood Cancer
MeSH Terms: conditions — Motor Activity; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical exercise program — At least two sessions a week for a 6-month supervised and individualized physical exercise program that will have two phases: one that will be carried out in person in the hospital environment taking advantage of medical visits, and a second phase that will allow the patient to carry out the exercise sessions from home with live virtual supervision.
Other: Type of the physical exercise program — Two types of intervention are proposed depending on the age of the patients: Exercise intervention for adolescents (12 to 18 years): training will be based on strength training (2 - 3 sets of 8 - 12 repetitions) with elastic bands, weights, weights, medicine balls or body weight and aerobic work on a stationary bike, treadmill or other aerobic exercises. Sessions will last about 30-60 minutes (depending on the patient's situation). Exercise intervention for children (4 to 11 years old): The aim will be to work on basic motor skills through play, thus trying to avoid the delay in motor development, and to indirectly work on their physical condition to better cope with the effects of the treatments. Music, games that require movement and materials such as balls, hoops, etc., will be used to motivate the child to move while enjoying themselves. This will be done in sessions of 20 - 40 minutes.

SUMMARY:
Objective: To assess the feasibility of a supervised, controlled and personalised physical exercise programme and its potential efficacy in improving functional capacity and quality of life in children and adolescents with cancer.

Design: Hybrid quasi-experimental pilot trial, clinical and phase I implementation.

Methods: The learning collaborative approach based on the Institute for Healthcare Improvement Breakthrough Series Collaborative Model will be followed through quarterly Plan-Do-Study-Act (P-D-S-A) cycles. Participants: For feasibility, at least, 45 patients will be included in 3 successive PDSA cycles of at least 15 patients each, aged 4-18 years diagnosed with any type of cancer. Variables: clinical and socio-demographic, body composition, physical condition and mobility, quality of life, physical activity and implementation. Intervention: Everyone will receive a physical exercise intervention combining strength and aerobic capacity work. Initially it will be carried out in the hospital setting, and later in streaming supervised by a professional. The intervention will be modelled through a formative evaluation process with the collaboration of all the agents involved, experimenting in each cycle with an increasingly adapted version of the exercise programme.

Statistical analysis: Recruitment rates will be calculated, characteristics associated with project participation and adherence to the exercise programme will be identified. Outcome variables will be compared before and after the intervention, identifying those with the greatest validity, reliability and sensitivity to change, which will then be used in phase II and III trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer and other neoplasms
* Age between 4 and 18 years at the time of inclusion in the study
* Patients diagnosed with cancer and other malignancies aged between 4 and 18 years who are experiencing relapse
* Paediatric patients requiring chemotherapy, radiotherapy, or oncological surgery
* Patients and parents or guardians who agree to participate in the study and sign the informed consent forms by current legislation depending on the patient's age.

Exclusion Criteria:

* Patients with cognitive deficits that prevent participation in and performance of physical exercise interventions.
* Patients with severe neurological pathology with a motor impairment that prevents or significantly hinders the performance of physical exercise
* Patients and families or guardians with language comprehension difficulties that make it difficult or impossible to carry out the physical exercise intervention.
* Patients < 16 years with a functional status score according to Lanskyi scale <60%
* Patients > 16 years with Karnofsky scale <60%.
* Any other criteria that the physician deems inappropriate for participation in the study

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Quarterly recruitment rates assessed by comparing those who participate with those who do not. | 2 years
  To assess the feasibility of the exercise programme, quarterly recruitment rates will be calculated over the recruitment and follow-up period, and socio-demographic and morbidity variables associated with study participation will be identified, comparing those who participate with those who do not, using logistic regression analysis.
Adherence rates assessed by the proportion of sessions completed and adherence to the prescribed exercise protocol | 2 years
  Participants' adherence to the programme will be described in terms of the proportion of sessions completed and compliance with the exercise protocol prescribed for each patient, and variables associated with compliance will be identified.
Body composition assessed by the Body Mass Index | 2 years
  Body Mass Index (BMI): Diagnoses and classifies obesity. weight and height will be combined to report BMI in kg/m^2). Measured at baseline, and 3 months.
Muscle mass | 3 months
  Muscle mass will be measured in kgs by a bioimpedance scale. Measured at baseline, and 3 months.
Bone mineral density | 3 months
  Bone mineral density will be in g/cm2 measured by a bioimpedance scale. Measured at baseline, and 3 months.
Physical condition assessed by the 6 min walking test and manual grip test with a dynamometer | 3 months
  The 6 minutes walking Test applies to assess functional capacity, as well as a predictor of morbidity and mortality in people with different pathologies. Most of the daily activities that the patients with these pathologies are performed at submaximal exercise intensity, similar to this test is performed. It would be measured at 0 and 3 months.
Muscular strength assessed by manual grip test with a dynamometer | 3 months
  The manual grip test with a dynamometer applies to assess muscular strength. Most of the daily activities that the patients with these pathologies are performed at submaximal exercise intensity, similar to this test is performed. It would be measured at 0 and 3 months.
General Quality of life assessed by the PedsQL 4.0 questionnaire | 3 months
  The PedsQL Measurement Model is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL Measurement Model integrates seamlessly both generic core scales and disease-specific modules into one measurement system. The questionnaire is self-reported for children over 8 years old and self-reported by parents for children under 8 years old. This questionnaire has been validated in the Spanish population. It would be measured at 0 and 3 months.
Specific Quality of life assessed by the PedsQL cancer questionnaire | 3 months
  The Pediatric Quality of Life Inventory (PedsQL) Cancer Module is a standard tool designed to assess the HRQOL among pediatric oncology patients. Consists of an instruction section and 27 items, contained in 8 dimensions. This questionnaire has been validated in the Spanish population. It would be measured at 0 and 3 months.
Fatigue assessed by the PedsQL Multidimensional Fatigue Scale Acute Version (PedsQL-MFS) | 3 months
  The PedsQL™ Multidimensional Fatigue Scale was designed as a generic symptom-specific instrument to measure fatigue in patients with acute and chronic health conditions as well as healthy school and community populations. The appropriate questionnaire will be used depending on the age of the patients (Toddlers (2-4 years of age), Young Child (5-7 years of age), Child (8-12 years of age), Adolescent (13-18 years of age)). This questionnaire has been validated in the Spanish population. It would be measured at 0 and 3 months.
Physical activity level assessed by accelerometers | 3 months
  Objectively registered with Actigraph wGT3X-BT accelerometer. Measured at 0 and 3 months

SECONDARY OUTCOMES:
Security assessment | 2 years
  To assess the safety of this new exercise programme by describing the occurrence of injuries, incidence of complications.
Costs associated estimation | 3 years
  Estimate the costs associated with the implementation of the programme.
Implementation barriers and facilitators | 2 years
  Describe the most important difficulties encountered in its implementation, identify barriers and facilitating factors for its implementation and realisation with minimum quality criteria, using the Consolidated Framework for Implementation Research (CFIR) as a theoretical framework for implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Menchaca Torio, Principal Investigator — Basque Health Service

IPD SHARING:
Plan to Share IPD: No